CLINICAL TRIAL: NCT03118869
Title: B2adrenergic Receptor Gene Polymorphism in Bronchial Asthma: Relation to Disease Severity and Control
Brief Title: B2 Adrenergic Receptor Gene Polymorphism in Bronchial Asthma
Acronym: polymorphism
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aliae AR Mohamed Hussein, Prof. Dr. Aliae AR Mohamed-Hussein, Professor of Pulmonology, Assiut University
Other Study IDs: AssiutU3
Record Dates: First submitted 2017-04-11; First posted 2017-04-18 (Actual); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Gene Abnormality; Asthma
Keywords: Asthma; B2 adrenergic receptors; Polymorphism
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The b2-adrenoceptor (b2AR) mediates the physiological responses in the airway, which include bronchodilation, bronchoprotection. The b2-adrenoceptor (b2AR) mediates the physiological responses in the airway, which include bronchodilation, bronchoprotection, Enhanced mucociliary clearance.

The b2AR gene is located on chromosome 5q31-q32, a region that is genetically linked to asthma and related phenotypes. There are three best known polymorphisms in the coding region of the b2AR gene that can modulate the function of the receptor.

DETAILED DESCRIPTION:
Asthma is a complex disease and has a strong genetic component in its pathogenesis. So far, considerable efforts have been made to evaluate the association between genetic variants and asthma risk, and numerous genes have been identified as asthma Reporting Items susceptible genes.

The b2-adrenoceptor (b2AR) mediates the physiological responses in the airway, which include bronchodilation, bronchoprotection. The b2-adrenoceptor (b2AR) mediates the physiological responses in the airway, which include bronchodilation, bronchoprotection, Enhanced mucociliary clearance.

The b2AR gene is located on chromosome 5q31-q32, a region that is genetically linked to asthma and related phenotypes. There are three best known polymorphisms in the coding region of the b2AR gene that can modulate the function of the receptor.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed as asthma according to GINA guideline 2016.
* Allergic asthma

Exclusion Criteria:

* pneumonia
* chronic cardiac, hepatic and renal diseases
* pregnancy and lactation
* malignancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed as asthma according to GINA 2016
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-10-01 (Estimated); Study Completion 2017-10-30 (Estimated)

PRIMARY OUTCOMES:
To measure number of patient with homozygous and heterozygous B2AD gene polymorphisms with focus on Arg/Gly16 and Gln/Glu27 polymorphism | 1 month
  study of prevalence homozygote and heterozygote patients

SECONDARY OUTCOMES:
Number of patient with b2AR gene polymorphisms in different asthma severity and different response of treatment of asthma ( Arg/Gly16 and Gln/Glu27 polymorphism) | 1 month
  correlation between polymorphism and pulmonary function test and level of disease control

CONTACTS AND LOCATIONS:
Overall Officials: Aliae Mohamed-Hussein, Principal Investigator — Professor of Pulmonology- Faculty of Medicine-Assiut University
Locations (1):
- AssiutU, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mohamed-Hussein AAR, Sayed SS, Eldien HMS, Assar AM, Yehia FE. Beta 2 Adrenergic Receptor Genetic Polymorphisms in Bronchial Asthma: Relationship to Disease Risk, Severity, and Treatment Response. Lung. 2018 Dec;196(6):673-680. doi: 10.1007/s00408-018-0153-3. Epub 2018 Sep 3. PMID 30178312